CLINICAL TRIAL: NCT00951470
Title: Lymphedema in Patients With Oral Cavity and Oropharyngeal Cancer: Prevalence, Functional Effects, and Treatment Outcomes
Brief Title: Complete Decongestive Therapy (CDT) for Treatment of Head and Neck Lymphedema
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0363
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Lymphedema; Oropharyngeal Cancer; Head and Neck Cancer; Oral Cancer
Keywords: Head and neck lymphedema; Complete Decongestive Therapy; CDT; Oral cavity cancer; Oropharyngeal cancer
MeSH Terms: conditions — Lymphedema; Oropharyngeal Neoplasms; Head and Neck Neoplasms; Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No CDT (Other): CDT=complete decongestive therapy
  Interventions: Other: Follow -Up Visits
- Modified CDT Program (Other): CDT=complete decongestive therapy
  Interventions: Other: Modified CDT Program
- Full CDT Program (Other): CDT=complete decongestive therapy
  Interventions: Other: Full CDT

INTERVENTIONS:
Other: Follow -Up Visits — If CDT is declined, participants will have follow-up visits at 1, 3, and 6 months after study interview.
  Arms: No CDT
Other: Full CDT — Monday through Friday visits to the clinic for 2 weeks of intensive outpatient therapy. The CDT will be done by the lymphedema therapist. Each session will last about 1 hour.
  During the last 2 treatment visits (Visits 9 and 10), the participant will be taught how to do the CDT steps at home. Then, the CDT steps will be performed at home, every day for the next 3 months.
  Other Names: complete decongestive therapy
  Arms: Full CDT Program
Other: Modified CDT Program — The participant will come to the clinic for 1-2 training sessions taught by the lymphedema therapist. Each training session will last about 1 hour, and the participant will be taught how to do the CDT steps at home. Then, the CDT steps will be performed at home, every day for the next 3 months.
  Other Names: complete decongestive therapy
  Arms: Modified CDT Program

SUMMARY:
Objectives:

Specific Aim 1: Estimate the prevalence of head and neck lymphedema in patients who have been treated with surgery and/or radiation therapy (± chemotherapy) for oral cavity and oropharyngeal cancer.

Compare functional outcomes in patients with and without lymphedema using cross-sectional survey methods.

Specific Aim 2: Evaluate the effect of Complete Decongestive Therapy (CDT) provided in an outpatient setting or a home-based program in reducing lymphedema in patients previously treated with surgery and/or radiation therapy (± chemotherapy) for oral cavity and oropharyngeal cancer at 1, 3 and 6 months follow-up. Patient characteristics, treatment variables, and the health care environment will be analyzed as possible explanatory variables that influence the effect of lymphedema treatment.

Specific Aim 3: Evaluate the effect of lymphedema treatment on symptom burden, self-image, and functional performance status in patients previously treated with surgery and/or radiation therapy (± chemotherapy) for oral cavity and oropharyngeal cancer.

DETAILED DESCRIPTION:
Screening for Part 1 of the Study:

The research staff will review your medical record to find out if you are possibly eligible to join Part 1 of this study. You will be eligible if you have had radiation and/or surgery (with or without chemotherapy) for mouth or throat cancer and it has been at least 1 month since your last treatment.

Part 1 of the Study:

If you choose to participate in Part 1 of this study, you will complete questionnaires. The questionnaires ask about your ability to swallow, eat, and speak, and about your quality of life, your satisfaction with your body, and any head and neck cancer symptoms. In total, the questionnaires should take less than 30 minutes to complete. You will also be asked about any symptoms of lymphedema. Your answers will be compared to the answers of patients who do and do not have lymphedema.

If you do not join Part 2 of this study, your participation in this study will be over after you complete the questionnaires.

Screening for Part 2 of the Study:

If you have head and neck lymphedema, you may also be eligible for Part 2 of the study. You will have "screening tests" to help the doctor decide if you are eligible for Part 2 of the study:

* The answers you provide to a questionnaire during Part 1 of the study will help the doctor find out if you may have lymphedema.
* Blood (about 1/2 teaspoon) will be drawn to check your thyroid function.
* Your doctor will also check your face and neck for signs of lymphedema during your regular clinic visit.

The research staff will discuss the Part 2 screening test results with you, if applicable. Signing this consent form does not mean that you will be able to participate in Part 2 of this study. If the screening tests show that you are not eligible for Part 2, you will only be enrolled in Part 1.

Part 2 of the Study:

If you are found to be eligible to take part in Part 2 of this study, you will first meet with a certified lymphedema therapist in the Head and Neck Center. During this visit, the therapist will perform a lymphedema exam. This involves checking your neck, face, and mouth for swelling, and looking at your skin to check for any open wounds or infection. The therapist will also interview you about how well you are able to swallow, eat, speak, and perform other normal activities of daily living (performance status). This visit should last about 1 hour.

All Part 2 participants will be offered CDT. It will be your choice if you would like to receive a "full" CDT program or a "modified" CDT program. You may also choose to decline both of these CDT options and stay on study for follow-up.

CDT has 4 steps that are designed to help the lymph fluids flow:

* Soft tissue of the face and neck is gently massaged, from inside or outside the mouth. This lasts for about 30-45 minutes.
* Bandages are placed on the face and neck in order to apply gentle pressure to the affected areas. The bandages stay in place for about 2-3 hours, before and/or after the massage.
* The face and neck muscles are exercised a certain way for about 15 minutes or less, while the bandages are in place.
* The face and neck is washed a certain way for about 5 minutes or less.

All 4 steps are done in both the full and modified CDT programs. The difference between the full and modified programs is that the full program includes 10 CDT sessions at the clinic, in addition to a self-managed CDT program at home. Otherwise, the 4 steps of CDT are the same in both the clinic sessions and home sessions.

Full CDT Program:

If you choose to receive the full CDT program, you will come to the clinic and receive CDT as described above, Monday through Friday for 2 weeks of intensive outpatient therapy. The CDT will be done by the lymphedema therapist. Each session will last about 1 hour.

During your last 2 treatment visits (Visits 9 and 10), you will be taught how to do the CDT steps at home. You will then perform the CDT steps at home, every day for the next 3 months.

Modified CDT Program:

If you choose to receive the modified CDT program, you will come to the clinic for 1-2 training sessions taught by the lymphedema therapist. Each training session will last about 1 hour, and you will be taught how to do the CDT steps at home. You will then perform the CDT steps at home, every day for the next 3 months.

Option for No CDT:

If you decline both study treatment options, you will not receive CDT. You will stay on study to receive follow-up as described below.

Follow-Up in Part 2 of the Study:

All Part 2 study participants will have 3 follow-up visits. If you received the full or modified CDT program, the visits will be at 1, 3, and 6 months after your first lymphedema training session. If you declined the CDT, the visits will be at 1, 3, and 6 months after your study interview.

At these visits, you will complete the same questionnaires as you did for screening in Part 1 of the study. You will also have a lymphedema exam and interview by the lymphedema therapist, like you did at the beginning of Part 2 of the study.

If you received the full or modified CDT program, a study staff member will also call you at 2, 6, and 9 weeks after your first lymphedema training session, to ask how the home CDT program is going.

Length of Part 2:

If you are in Part 2, your participation in this study will be over after your 6-month follow-up visit.

This is an investigational study. CDT is commonly used to treat all types of lymphedema, including head and neck lymphedema. This study (Part 2) is designed to collect more data on whether CDT can help to control head and neck lymphedema and its symptoms. Part 1 is also designed to collect data related to head and neck lymphedema.

Up to 500 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (greater than or equal to 18 years of age) patients previously treated with definitive surgical resection and/or radiation therapy with or without chemotherapy for oral and/or oropharyngeal cancer who are at least 1 month posttreatment will be eligible for enrollment.
2. Patients who meet the above requirement and are also diagnosed with head and neck lymphedema by their physician will be eligible for participation in the prospective phase of the study.
3. Patients will be free of acute tissue reactions including oral mucositis, skin breakdown, and fistula prior to inclusion in the prospective phase of the study.
4. Patients will have baseline Thyroid Stimulating Hormone testing prior to inclusion in the prospective phase of the study.

Exclusion Criteria:

1. Patients who are actively being treated for head and neck cancer.
2. Patients whose cancer treatment was administered with palliative intent.
3. Patients with recurrent or second primary head and neck cancer, or persistent disease. Patients who have a persistent neck mass at completion of primary radiotherapy that necessitates salvage neck dissection will be ineligible for enrollment until 1 month (6 weeks) following neck dissection.
4. Patients with any of the following contraindications to lymphedema therapy: acute infection, active cancer, congestive heart failure, renal failure, cardiac or pulmonary edema, sensitive carotid sinus, severe carotid blockage, and uncontrolled hypertension.
5. Patients with edema related to hypothyroidism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Head & Neck Lymphedema Occurence | 30 minutes to complete questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jan S Lewin, PhD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org